CLINICAL TRIAL: NCT06921577
Title: Microbial and Laboratory Study of 3D Printed Reinforced Acrylic Denture
Brief Title: Clinical and Microbial Study of Reinforced 3D Printed Maxillary Denture Base Resin
Acronym: dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Teama, assistant lecturere in prosthodontics departement faculty of dentistry Tanta univrtsity, Tanta University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: RP 2-23 1
Record Dates: First submitted 2025-03-14; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Denture Stomatitis
Keywords: 3Dprinted resin; nanoparticles; antimicrobial effect
MeSH Terms: conditions — Stomatitis, Denture | interventions — Anti-Infective Agents

STUDY DESIGN:
Intervention Model Description: This study aimed to compare the effects of adding nanoZrO2 (0.4% wt) and nanoTiO2 (0.4% wt) to 3D-printed acrylic resin dentures in complete edentulous patients on microbial colonization and patient satisfaction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nanoparticles (Experimental): Group II: Patients used maxillary complete dentures 3D after reinforcement by Nano-ZrO2 (0.4%) by Wt. Group III: Patients used maxillary complete dentures 3D printed after reinforcement by Nano-TiO2 (0.4%) by Wt
  Interventions: Combination Product: antimicrobial agent

INTERVENTIONS:
Combination Product: antimicrobial agent — Adding nanoparticles to 3Dprinted denture base resin improve the properties of the material
  Other Names: antimcrobial ffect

SUMMARY:
Statement of problem: 3D printed denture base resin is needed to reinforce Purpose: To evaluate the effects of adding nano-ZrO2 and nano-TiO2 on microbial colonization and patient satisfaction with 3D-printed maxillary complete dentures.

Materials and Methods: Twenty-four patients who needed complete dentures were randomly distributed into three equal groups. Group I: Patients used maxillary complete dentures 3D printed without additives. Group II: Patients used maxillary complete dentures 3D after reinforcement by Nano-ZrO2 (0.4%) by Wt. Group III: Patients used maxillary complete dentures 3D printed after reinforcement by Nano-TiO2 (0.4%) by Wt. For microbial evaluation, a cotton swab was taken from the mucosa and the intaglio surface of maxillary dentures, and microbial colonization was evaluated by calculating the number of colony-forming units of S. aureus on mannitol salt agar plates and C. albicans on Sabouraud's dextrose agar plates after 48 hours of incubation at insertion, 6 months, 12 months and 18 months. Patient satisfaction was evaluated 15 days after insertion and at 6, 12, and 18 months. The values of microbial colonization and patient satisfaction were analyzed via repeated-measures ANOVA followed by Tukey's multiple comparison test.

DETAILED DESCRIPTION:
This study aims to compare the effect of 3D printed denture base without nanoparticles and 3D printed denture base reinforced with ZrO2 and TiO2 nanoparticles on completely edentulous patients, as regards:

1. Microbial colonization.
2. Patient satisfaction.

The following steps will be carried out for all patients:

1. Conventional primary and final impressions will be made for each patient
2. Master casts (upper and lower) and occlusion blocks will be scanned by an extra-oral scanner.
3. Files in standard tessellation language (STL) format of master casts and jaw relation records will be imported to the software platform. The software will enable virtually simultaneous mounting and aligning. Each denture will have two STL files that will be printed separately: one for the denture base and one for the teeth, using a 3D printer.29
4. For Group Ι, the designed dentures STL files will be sent to the 3D printer software. Pink denture base resin will be used to print denture bases without nanoparticles.
5. For Group II, Pink denture base resin reinforced by Nanoparticles (ZrO2) will be used to print denture bases.
6. For Group Ш, Pink denture base resin reinforced by Nanoparticles (TiO2) will be used to print denture bases.
7. White teeth resin will be utilized for teeth printing for all groups. Finally, teeth will be attached to recessed pockets in the dentures bases via resin. Followed by finishing. Eventually, dentures will be placed in the post-curing unit.

All patients will be given similar post insertion instructions and a regular oral and denture hygiene protocol.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients with good local and systemic health.
* Patients' ages range from 50 to 70 years old.
* Must have adequate interarch space and class Ⅰ angle classification.
* Must have a reasonable neuromuscular control. Patient exclusion criteria
* Patients with any diseases that may affect denture construction
* Patients with oral parafunctional habits.
* Patients with tempromandibular disorders

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Antimicrobial effect | 18 months
  Cotton swabs were taken from the mucosa and the intaglio surface of maxillary dentures, and microbial colonization was evaluated by calculating the number of colony-forming units of S. aureus on mannitol salt agar plates and C. albicans on Sabouraud's dextrose agar plates after 48 hours of incubation at insertion, 6 months, 12 months and 18 months.
Patient satisfaction | 18 months
  Patient satisfaction was evaluated 15 days after insertion and at 6, 12, and 18 months. Patients were requested to assess their overall satisfaction with their dentures through the visual analog scale. The patients were asked five questions: "How satisfied were you with your prosthesis considering aesthetics, speech, masticatory efficiency, hygiene, and comfort?" A ten-point scale was used to evaluate each question; the minimum score is zero, while the maximum score is ten. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Houda MA Rashad, professor, Study Director — Tanta University
Locations (1):
- Faculty of dentistry Tanta university Egypt, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
According to the guidelines of human research adopted by the Research Ethics Committee, Faculty of Dentistry, Tanta University.

REFERENCES:
- [Derived] Ahmed Teama EM, Amin Rashad HM, Mohamed Shakal EAE, Hegazy EE. Clinical and microbial study of reinforced 3D-printed maxillary denture base resin: a randomized trial. BMC Oral Health. 2025 Jul 17;25(1):1192. doi: 10.1186/s12903-025-06601-2. PMID 40676540